CLINICAL TRIAL: NCT01658878
Title: A Phase 1/2, Dose-escalation, Open-label, Non-comparative Study of Nivolumab or Nivolumab in Combination With Ipilimumab in Advanced Hepatocellular Carcinoma Subjects With or Without Chronic Viral Hepatitis; and a Randomized, Open-label Study of Nivolumab vs Sorafenib in Advanced Hepatocellular Carcinoma Subjects Who Are Naive to Systemic Therapy
Brief Title: An Immuno-therapy Study to Evaluate the Effectiveness, Safety and Tolerability of Nivolumab or Nivolumab in Combination With Other Agents in Patients With Advanced Liver Cancer
Acronym: CheckMate040
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-040; 2012-001514-42 (EudraCT Number)
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Sorafenib; Ipilimumab; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Non-infected: Nivolumab (Experimental): Nivolumab intravenous solution on specific days
  Interventions: Biological: Nivolumab
- HCV-infected: Nivolumab (Experimental): Nivolumab intravenous solution on specific days
  Interventions: Biological: Nivolumab
- HBV-infected: Nivolumab (Experimental): Nivolumab intravenous solution on specific days
  Interventions: Biological: Nivolumab
- Nivolumab (Experimental): Nivolumab intravenous solution on specific days
  Interventions: Biological: Nivolumab
- Sorafenib (Active Comparator): Sorafenib tablets on specific days
  Interventions: Drug: Sorafenib
- Nivolumab plus Ipilimumab Combination (Experimental): Nivolumab intravenous solution + Ipilimumab intravenous solution on specific days
  Interventions: Biological: Nivolumab; Drug: Ipilimumab
- Child-Pugh B (Experimental): Nivolumab intravenous solution on specific days
  Interventions: Biological: Nivolumab
- Nivolumab plus Cabozantinib Combination (Experimental): Nivolumab intravenous solution + cabozantinib oral tablets on specific days
  Interventions: Drug: Cabozantinib
- Nivolumab plus Ipilimumab plus Cabozantinib (Experimental): Nivolumab intravenous solution + Ipilimumab intravenous solution + cabozantinib oral tablets on specific days
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558
  Arms: Child-Pugh B; HBV-infected: Nivolumab; HCV-infected: Nivolumab; Nivolumab; Nivolumab plus Ipilimumab Combination; Non-infected: Nivolumab
Drug: Sorafenib
  Arms: Sorafenib
Drug: Ipilimumab
  Arms: Nivolumab plus Ipilimumab Combination
Drug: Cabozantinib
  Arms: Nivolumab plus Cabozantinib Combination; Nivolumab plus Ipilimumab plus Cabozantinib

SUMMARY:
The first part of the study is the Dose Escalation Phase designed to establish the safety of nivolumab at different dose levels for each of the three cohorts (uninfected hepatocellular carcinoma (HCC) subjects, hepatitis C virus (HCV)-infected HCC subjects, and hepatitis B virus (HBV)-infected subjects).

The second part of the study is the Expansion Phase designed to generate additional clinical data at specified doses for each of the 3 cohorts. A third cohort has been added in this study to compare the efficacy of nivolumab and sorafenib in the treatment of Advanced HCC. A fourth cohort will generate data on the safety and efficacy of the combination nivolumab plus ipilimumab in the treatment of Advanced HCC. In the fifth cohort, additional clinical data will be generated for Child-Pugh B subjects. A Cabozantinib Combination Cohort has been added to evaluate the safety and tolerability of nivolumab in combination with cabozantinib and nivolumab with ipilimumab in combination with cabozantinib.

DETAILED DESCRIPTION:
Study Classification: Pharmacokinetics/Pharmacodynamics

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects of 18 years or older (men and women) with histologically confirmed advanced hepatocellular carcinoma, not eligible for surgical and/or locoregional therapies; or progressive disease after surgical and /or locoregional therapies
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Dose Escalation Phase: Child-Pugh score of 7 points or less. Cohort 5: Child-Pugh Class B (B7-B8). For all other cohorts Child-Pugh score of 6 points or less

Exclusion Criteria:

* History of autoimmune disease
* Any prior or current clinically significant ascites
* Any history of hepatic encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (10):
  - Local Institution - 0008, Los Angeles, California
  - Local Institution - 0048, Washington D.C., District of Columbia
  - Local Institution - 0053, Pensacola, Florida
  - Local Institution - 0047, Atlanta, Georgia
  - Local Institution - 0025, Boston, Massachusetts
  - Local Institution - 0002, Ann Arbor, Michigan
  - Local Institution - 0054, Hackensack, New Jersey
  - Local Institution - 0067, Paterson, New Jersey
  - Local Institution - 0001, Portland, Oregon
  - The University Of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (3):
  - Local Institution - 0065, Halifax, Nova Scotia
  - Local Institution - 0039, Toronto, Ontario
  - Local Institution - 0022, Montreal, Quebec
- France (7):
  - Local Institution - 0061, Angers
  - Local Institution - 0064, Créteil
  - Local Institution - 0062, Marseille
  - Local Institution - 0059, Marseille
  - Local Institution - 0042, Paris
  - Local Institution - 0060, Reims
  - Local Institution - 0058, Vandœuvre-lès-Nancy
- Germany (4):
  - Local Institution - 0030, Essen
  - Local Institution - 0028, Frankfurt
  - Local Institution - 0029, Hanover
  - Local Institution - 0031, Heidelberg
- Hong Kong (2):
  - Local Institution - 0005, Hong Kong
  - Local Institution - 0006, Hong Kong
- Italy (7):
  - Local Institution - 0032, Bologna
  - Local Institution - 0056, Florence
  - Local Institution - 0063, Meldola (FC)
  - Local Institution - 0055, Milan
  - Local Institution - 0034, Napoli
  - Local Institution - 0035, Padua
  - Local Institution - 0040, Rozzano
- Japan (6):
  - Local Institution - 0036, Kashiwa-shi, Chiba
  - Local Institution - 0038, Kurume-shi, Fukuoka
  - Local Institution - 0049, Yokohama, Kanagawa
  - Local Institution - 0050, Kyoto, Kyoto
  - Local Institution - 0037, Ōsaka-sayama, Osaka
  - Local Institution - 0051, Saga
- Local Institution - 0070, San Juan, Puerto Rico
- Singapore (3):
  - Local Institution - 0017, Singapore
  - Local Institution - 0009, Singapore
  - Local Institution - 0007, Singapore
- South Korea (4):
  - Local Institution - 0066, Seoul
  - Local Institution - 0021, Seoul
  - Local Institution - 0026, Seoul
  - Local Institution - 0016, Seoul
- Spain (4):
  - Local Institution - 0019, Barcelona
  - Local Institution - 0020, Madrid
  - Local Institution - 0018, Madrid
  - Local Institution - 0003, Pamplona
- Taiwan (3):
  - Local Institution - 0027, Taipei
  - Local Institution - 0024, Taipei
  - Local Institution - 0023, Taoyuan District
- United Kingdom (6):
  - Local Institution - 0011, London, Greater London
  - Local Institution - 0014, Manchester, Greater Manchester
  - Local Institution - 0012, Glasgow, Lanarkshire
  - Local Institution - 0015, Metropolitan Borough of Wirral, Merseyside
  - Local Institution - 0013, Birmingham, West Midlands
  - Local Institution - 0010, London

REFERENCES:
- [Derived] Zhou X, Cao J, Topatana W, Xie T, Chen T, Hu J, Li S, Juengpanic S, Lu Z, Zhang B, Wang K, Feng X, Shen J, Chen M. Evaluation of PD-L1 as a biomarker for immunotherapy for hepatocellular carcinoma: systematic review and meta-analysis. Immunotherapy. 2023 Apr;15(5):353-365. doi: 10.2217/imt-2022-0168. Epub 2023 Feb 27. PMID 36852452
- [Derived] Yau T, Zagonel V, Santoro A, Acosta-Rivera M, Choo SP, Matilla A, He AR, Cubillo Gracian A, El-Khoueiry AB, Sangro B, Eldawy TE, Bruix J, Frassineti GL, Vaccaro GM, Tschaika M, Scheffold C, Koopmans P, Neely J, Piscaglia F. Nivolumab Plus Cabozantinib With or Without Ipilimumab for Advanced Hepatocellular Carcinoma: Results From Cohort 6 of the CheckMate 040 Trial. J Clin Oncol. 2023 Mar 20;41(9):1747-1757. doi: 10.1200/JCO.22.00972. Epub 2022 Dec 13. PMID 36512738
- [Derived] Sove RJ, Verma BK, Wang H, Ho WJ, Yarchoan M, Popel AS. Virtual clinical trials of anti-PD-1 and anti-CTLA-4 immunotherapy in advanced hepatocellular carcinoma using a quantitative systems pharmacology model. J Immunother Cancer. 2022 Nov;10(11):e005414. doi: 10.1136/jitc-2022-005414. PMID 36323435
- [Derived] Kudo M, Matilla A, Santoro A, Melero I, Gracian AC, Acosta-Rivera M, Choo SP, El-Khoueiry AB, Kuromatsu R, El-Rayes B, Numata K, Itoh Y, Di Costanzo F, Crysler O, Reig M, Shen Y, Neely J, Tschaika M, Wisniewski T, Sangro B. CheckMate 040 cohort 5: A phase I/II study of nivolumab in patients with advanced hepatocellular carcinoma and Child-Pugh B cirrhosis. J Hepatol. 2021 Sep;75(3):600-609. doi: 10.1016/j.jhep.2021.04.047. Epub 2021 May 26. PMID 34051329
- [Derived] Yau T, Kang YK, Kim TY, El-Khoueiry AB, Santoro A, Sangro B, Melero I, Kudo M, Hou MM, Matilla A, Tovoli F, Knox JJ, Ruth He A, El-Rayes BF, Acosta-Rivera M, Lim HY, Neely J, Shen Y, Wisniewski T, Anderson J, Hsu C. Efficacy and Safety of Nivolumab Plus Ipilimumab in Patients With Advanced Hepatocellular Carcinoma Previously Treated With Sorafenib: The CheckMate 040 Randomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):e204564. doi: 10.1001/jamaoncol.2020.4564. Epub 2020 Nov 12. PMID 33001135
- [Derived] Sangro B, Melero I, Wadhawan S, Finn RS, Abou-Alfa GK, Cheng AL, Yau T, Furuse J, Park JW, Boyd Z, Tang HT, Shen Y, Tschaika M, Neely J, El-Khoueiry A. Association of inflammatory biomarkers with clinical outcomes in nivolumab-treated patients with advanced hepatocellular carcinoma. J Hepatol. 2020 Dec;73(6):1460-1469. doi: 10.1016/j.jhep.2020.07.026. Epub 2020 Jul 22. PMID 32710922
- [Derived] Yau T, Hsu C, Kim TY, Choo SP, Kang YK, Hou MM, Numata K, Yeo W, Chopra A, Ikeda M, Kuromatsu R, Moriguchi M, Chao Y, Zhao H, Anderson J, Cruz CD, Kudo M. Nivolumab in advanced hepatocellular carcinoma: Sorafenib-experienced Asian cohort analysis. J Hepatol. 2019 Sep;71(3):543-552. doi: 10.1016/j.jhep.2019.05.014. Epub 2019 Jun 7. PMID 31176752
- [Derived] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 657 participants were randomized and 650 received treatment across six cohorts. Randomization occurred in Cohorts 3, 4, and 6, while Cohorts 1, 2, and 5 included non-randomized participants.
Groups:
- Cohort 1 Uninfected HCC: Treatment 1: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 0.1 mg/kg every 2 weeks
- Cohort 1 Uninfected HCC: Treatment 2: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 0.3 mg/kg every 2 weeks
- Cohort 1 Uninfected HCC: Treatment 3: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 1 mg/kg every 2 weeks
- Cohort 1 Uninfected HCC: Treatment 4: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 3 mg/kg every 2 weeks
- Cohort 1 Uninfected HCC: Treatment 5: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 10 mg/kg every 2 weeks
- Cohort 1 HCV Infected: Treatment 6: Dose Escalation: Hepatitis C (HCV)-infected participants received nivolumab 0.3 mg/kg every 2 weeks
- Cohort 1 HCV Infected: Treatment 7: Dose Escalation: Hepatitis C (HCV)-infected participants received nivolumab 1 mg/kg every 2 weeks
- Cohort 1 HCV Infected: Treatment 8: Dose Escalation: Hepatitis C (HCV)-infected participants received nivolumab 3 mg/kg every 2 weeks
- Cohort 1 HBV Infected: Treatment 9: Dose Escalation: Hepatitis B (HBV)-infected participants received nivolumab 0.1 mg/kg every 2 weeks
- Cohort 1 HBV Infected: Treatment 10: Dose Escalation: Hepatitis B (HBV)-infected participants received nivolumab 0.3 mg/kg every 2 weeks
- Cohort 1 HBV Infected: Treatment 11: Dose Escalation: Hepatitis B (HBV)-infected participants received nivolumab 1 mg/kg every 2 weeks
- Cohort 1 HBV Infected: Treatment 12: Dose Escalation: Hepatitis B (HBV)-infected participants received nivolumab 3 mg/kg every 2 weeks
- Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1: Dose Expansion: Uninfected hepatocellular carcinoma (HCC) participants who are sorafenib naive/intolerant received nivolumab 3 mg/kg every 2 weeks
- Cohort 2 Uninfected Sorafenib Progressors: Treatment 2: Dose Expansion: Uninfected hepatocellular carcinoma (HCC) participants who are sorafenib progressors received nivolumab 3 mg/kg every 2 weeks
- Cohort 2 HCV Infected: Treatment 3: Dose Expansion: Hepatitis C (HCV)-infected participants received nivolumab 3 mg/kg every 2 weeks
- Cohort 2 HBV Infected: Treatment 4: Dose Expansion: Hepatitis B (HBV)-infected participants received nivolumab 3 mg/kg every 2 weeks
- Cohort 3: Treatment 1: Arm A: Advance hepatocellular carcinoma (HCC) participants received nivolumab 240 mg every 2 weeks
- Cohort 3: Treatment 2: Arm B: Advance hepatocellular carcinoma (HCC) participants received Sorafenib 400 mg twice a day
- Cohort 4: Treatment 1: Arm A: Participants received nivolumab 1 mg/kg + ipilimumab 3 mg/kg every 3 weeks
- Cohort 4: Treatment 2: Arm B: Participants received nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks
- Cohort 4: Treatment 3: Arm C: Participants received nivolumab 3 mg/kg every 2 weeks + ipilimumab 1 mg/kg every 6 weeks
- Cohort 5: Treatment 1: Participants received nivolumab 240 mg every 2 weeks
- Cohort 6: Treatment 1: Participants received nivolumab 240 mg every 2 weeks + cabozantinib 40 mg once daily
- Cohort 6: Treatment 2: Participants received nivolumab 3 mg/kg every 2 weeks + ipilimumab 1 mg/kg every 6 weeks + cabozantinib 40 mg once daily
Period: Pre-Treatment Period
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Started | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Randomized | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 66 | 50 | 49 | 49 | 0 | 36 | 35
Completed (Completed = Moved to treatment period) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Started (Started = Treated) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Not completed — Disease Progression | 1 | 3 | 2 | 1 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 43 | 48 | 33 | 46 | 41 | 42 | 28 | 37 | 37 | 39 | 27 | 19
Not completed — Study Drug Toxicity | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 5 | 0 | 5 | 10 | 12 | 4 | 2 | 3 | 2 | 6
Not completed — Maximum Clinical Benefit | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 3 | 1 | 4 | 0 | 0 | 4
Not completed — Participant No Longer Meets Study Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Poor/Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 2
Not completed — Participant Request to Discontinue Study Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 2 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 1
Not completed — Adverse Event Related to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 3 | 3 | 2 | 3 | 3 | 4 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2 | Total
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35 | 657
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 2 | 9 | 2 | 2 | 0 | 1 | 2 | 3 | 3 | 23 | 28 | 25 | 38 | 24 | 33 | 31 | 24 | 36 | 16 | 18 | 16 | 340
  >=65 years | 0 | 1 | 2 | 1 | 4 | 1 | 2 | 3 | 4 | 1 | 0 | 1 | 33 | 29 | 25 | 13 | 37 | 33 | 19 | 25 | 13 | 33 | 18 | 19 | 317
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 8 | 15 | 8 | 12 | 10 | 10 | 7 | 12 | 9 | 10 | 4 | 5 | 122
  Male | 1 | 1 | 3 | 2 | 10 | 2 | 3 | 1 | 4 | 3 | 2 | 4 | 48 | 42 | 42 | 39 | 51 | 56 | 43 | 37 | 40 | 39 | 32 | 30 | 535
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 2 | 3 | 3 | 11 | 3 | 3 | 2 | 1 | 0 | 0 | 0 | 38 | 34 | 29 | 4 | 39 | 42 | 12 | 20 | 15 | 27 | 26 | 23 | 337
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 1 | 3 | 2 | 2 | 1 | 21
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4 | 3 | 3 | 4 | 16 | 22 | 18 | 45 | 19 | 21 | 37 | 27 | 30 | 20 | 8 | 10 | 291
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 6
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose of study medication through 100 days following last dose of study treatment (Assessed approximately 04 months up to a max of approximately 106 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Participants | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 56 | 50 | 51 | 58 | 59 | 48 | 47 | 48 | 47 | 36 | 35

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, and requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: as for outcome 1
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Participants | 0 | 1 | 2 | 0 | 5 | 0 | 3 | 1 | 5 | 3 | 0 | 2 | 34 | 28 | 29 | 21 | 27 | 25 | 30 | 27 | 29 | 31 | 17 | 21

3. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Participants | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 8 | 10 | 3 | 14 | 16 | 16 | 7 | 10 | 8 | 7 | 12

4. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died during the study.
Time Frame: From first dose of study medication until study closure (Up to approximately 144 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 50 | 51 | 60 | 62 | 49 | 49 | 48 | 49 | 36 | 35
Participants | 1 | 3 | 2 | 2 | 13 | 1 | 4 | 3 | 5 | 3 | 3 | 4 | 49 | 52 | 40 | 45 | 52 | 53 | 35 | 41 | 40 | 48 | 29 | 26

5. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Participants with abnormalities in liver function tests related to potential drug-induced liver injury. Blood samples were collected and analyzed for liver function parameters, including alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Abnormalities were assessed relative to the upper limit of normal (ULN) for each parameter.
  Abbreviations: ALT = Alanine Aminotransferase; AST = Aspartate Aminotransferase; ULN = Upper Limit of Normal.
Time Frame: as for outcome 1
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 57 | 48 | 51 | 59 | 60 | 47 | 49 | 45 | 47 | 35 | 34
Participants
  ALT or AST > 3 X Upper limit of Normal (ULN) | 0 | 1 | 1 | 1 | 7 | 2 | 4 | 1 | 2 | 0 | 2 | 2 | 22 | 20 | 32 | 12 | 23 | 21 | 29 | 25 | 23 | 27 | 23 | 21
  Alanine Transaminase (ALT) OR AST > 5 X ULN | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 1 | 2 | 0 | 2 | 1 | 10 | 10 | 22 | 5 | 9 | 7 | 22 | 14 | 11 | 17 | 12 | 19
  ALT or Aspartate Transaminase (AST) > 10 X ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 5 | 10 | 4 | 3 | 2 | 8 | 7 | 7 | 2 | 5 | 9
  ALT or AST > 15 X ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 3 | 1 | 3 | 2 | 2 | 3 | 2 | 1 | 1 | 3
  ALT or AST > 20 X ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 2
  Total Bilirubin > 2 X ULN | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 5 | 9 | 10 | 6 | 13 | 12 | 11 | 9 | 2 | 17 | 5 | 8
  Total Bilirubin > 8 X ULN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3 | 0 | 5 | 4 | 0 | 1 | 0 | 1
  Total Bilirubin >8XULN if Elevated at Entry Or >5XULN if Normal at Entry | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 3 | 0 | 5 | 4 | 0 | 2 | 0 | 1
  Concurrent ALT OR AST Elevation > 3 X ULN with Total Bilirubin > 2 X ULN within One Day | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 6 | 7 | 5 | 9 | 10 | 9 | 7 | 1 | 10 | 4 | 7
  Concurrent ALT or AST elevation > 3 X ULN with Total Bilirubin > 2 X ULN within 30 Days | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3 | 6 | 7 | 5 | 9 | 11 | 9 | 7 | 1 | 11 | 4 | 7
  Concurrent Alt>=10XULN & Total Bilirubin >=2XULN Or 2X Baseline if Elevated Total Bilirubin at Entry | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants with thyroid-related laboratory abnormalities during the study. Blood samples were collected and analyzed for thyroid function markers (FT3, FT4). Abnormalities were assessed against LLN and ULN for each parameter.
  Abbreviations: FT3 = Free T3; FT4 = Free T4; LLN = Lower Limit of Normal; ULN = Upper Limit of Normal; TSH = Thyroid Stimulating Hormone
Time Frame: as for outcome 1
Population: All treated participants with at least one on-treatment thyroid stimulating hormone (TSH) measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 13 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 56 | 56 | 47 | 50 | 54 | 57 | 41 | 38 | 42 | 41 | 35 | 32
Participants
  TSH > ULN (Upper Limit of Normal) | 0 | 1 | 1 | 1 | 5 | 1 | 1 | 3 | 0 | 1 | 0 | 1 | 20 | 23 | 21 | 17 | 15 | 19 | 23 | 15 | 15 | 6 | 21 | 17
  TSH > ULN with TSH <= ULN at baseline | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 15 | 17 | 13 | 11 | 11 | 15 | 18 | 11 | 9 | 5 | 20 | 14
  TSH > ULN with at least one FT3/FT4 test value < LLN (Lower Limit of Normal) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 7 | 14 | 6 | 5 | 6 | 6 | 10 | 8 | 4 | 3 | 6 | 7
  TSH > ULN with all other FT3/FT4 test values >= LLN | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 11 | 8 | 14 | 10 | 6 | 9 | 11 | 4 | 5 | 3 | 11 | 6
  TSH > ULN with FT3/FT4 test missing | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 3 | 4 | 2 | 3 | 6 | 0 | 4 | 4
  TSH < LLN | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 10 | 7 | 8 | 9 | 2 | 6 | 16 | 13 | 10 | 5 | 6 | 9
  TSH < LLN with TSH >= LLN at baseline | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 7 | 7 | 7 | 2 | 4 | 15 | 12 | 9 | 5 | 4 | 9
  TSH < LLN with at least one FT3/FT4 test value > ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 3 | 4 | 1 | 1 | 2 | 9 | 6 | 6 | 2 | 2 | 5
  TSH < LLN with all other FT3/FT4 test values <= ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 3 | 8 | 1 | 4 | 5 | 2 | 3 | 1 | 3 | 4
  TSH < LLN with FT3/FT4 test missing | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 1 | 2 | 1 | 0

7. Primary Outcome: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) for Cohort 2
Description: Objective response rate (ORR) is defined as the percent of all treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) by BICR per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the start of the study treatment until disease progression, or the date of subsequent anti-cancer therapy, whichever occurs first (Up to approximately 144 months)
Population: All treated participants for Cohort 2 only. Pre-specified to be reported for Cohort 2 only.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4
Number analyzed (Participants) | 56 | 57 | 50 | 51
Percent of Participants | 19.6 [10.2 to 32.4] | 14.0 [6.3 to 25.8] | 20.0 [10.0 to 33.7] | 13.7 [5.7 to 26.3]

8. Primary Outcome: Objective Response Rate (ORR) by Investigator for Cohorts 3, 4, 5, and 6
Description: Objective response rate (ORR) is defined as the percent of all treated participants whose best overall response (BOR) is either complete response (CR) or partial response (PR) by Investigator per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 5) until disease progression, or the date of subsequent anti-cancer therapy, whichever occurs first (Up to approximately 144 months)
Population: All treated participants for Cohorts 05, and all randomized participants for Cohorts 03, 04 and 06 only. Pre-specified to be reported for Cohorts 3 through 6.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Percent of Participants | 11.5 [4.7 to 22.2] | 4.5 [0.9 to 12.7] | 36.0 [22.9 to 50.8] | 26.5 [14.9 to 41.1] | 28.6 [16.6 to 43.3] | 12.2 [4.6 to 24.8] | 16.7 [6.4 to 32.8] | 25.7 [12.5 to 43.3]

9. Secondary Outcome: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review (BICR) for Cohort 1
Description: as for outcome 7
Time Frame: as for outcome 7
Population: All treated participants in Cohort 1; uninfected HCC, HCV-infected, and HBV-infected participants reported together as pre-specified.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Cohort 1 Uninfected HCC: Dose Escalation: Uninfected hepatocellular carcinoma (HCC) participants received nivolumab 0.1/0.3/1/3/10 mg/kg every 2 weeks
- Cohort 1 HCV Infected: Dose Escalation: Hepatitis C (HCV)-infected participants received nivolumab 0.3/1/3 mg/kg every 2 weeks
- Cohort 1 HBV Infected: Dose Escalation: Hepatitis B (HBV)-infected participants received nivolumab 0.1/0.3/1/3 mg/kg every 2 weeks
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 23 | 10 | 15
Percent of Participants | 13.0 [2.8 to 33.6] | 20.0 [2.5 to 55.6] | 13.3 [1.7 to 40.5]

10. Secondary Outcome: Number of Participants With Complete Response (CR) Assessed by Blinded Independent Central Review (BICR)
Description: The number of participants whose best overall response (BOR) is CR in the population of interest. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) up to approximately 144 months after first dose
Population: All treated participants for Cohort 1, 2, and 5, and all randomized participants for Cohort 3, 4 and 6. Uninfected HCC, HCV-infected, and HBV-infected participants were pre-specified to be reported together for Cohort 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Participants | 1 | 0 | 0 | 2 | 0 | 2 | 4 | 1 | 1 | 4 | 4 | 1 | 0 | 1 | 3

11. Secondary Outcome: Disease Control Rate (DCR) Assessed by Blinded Independent Central Review (BICR)
Description: The percentage of participants whose best overall response (BOR) is CR, PR or SD in the population of interest. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Failure to meet criteria for complete or partial response, in the absence of progressive disease. Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) until disease progression, or the date of subsequent anti-cancer therapy, whichever occurs first (Up to approximately 144 months)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Percent of Participants | 47.8 [26.8 to 69.4] | 70.0 [34.8 to 93.3] | 40.0 [16.3 to 67.7] | 66.1 [52.2 to 78.2] | 56.1 [42.4 to 69.3] | 54.0 [39.3 to 68.2] | 47.1 [32.9 to 61.5] | 52.5 [39.3 to 65.4] | 62.1 [49.3 to 73.8] | 54.0 [39.3 to 68.2] | 42.9 [28.8 to 57.8] | 49.0 [34.4 to 63.7] | 44.9 [30.7 to 59.8] | 77.8 [60.8 to 89.9] | 80.0 [63.1 to 91.6]

12. Secondary Outcome: Duration of Response (DOR) Assessed by Blinded Independent Central Review (BICR)
Description: DOR is defined as the time from the first documented objective response (either complete or partial response) until the date of disease progression or death from any cause, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From first documented response to first documented progression or death, whichever occurs first (Up to approximately 144 months)
Population: All treated participants for Cohort 1, 2, and 5, and all randomized participants for Cohort 3, 4 and 6 whose best overall response (BOR) is either complete response (CR) or partial response (PR). Uninfected HCC, HCV-infected, and HBV-infected participants were pre-specified to be reported together for Cohort 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 3 | 2 | 2 | 11 | 8 | 10 | 7 | 8 | 4 | 16 | 16 | 15 | 3 | 5 | 10
Months | NA [8.74 to NA] — Not estimable due to insufficient number of events | 12.55 [5.75 to NA] — Insufficient number of events to calculate UL | 6.41 [2.83 to NA] — Insufficient number of events to calculate UL | 22.57 [5.62 to 31.80] | 11.30 [5.55 to NA] — Insufficient number of events to calculate UL | NA [3.15 to NA] — Not estimable due to insufficient number of events | NA [8.31 to NA] — Not estimable due to insufficient number of events | 5.21 [2.10 to NA] — Insufficient number of events to calculate UL | 9.26 [5.45 to NA] — Insufficient number of events to calculate UL | 17.48 [8.31 to 52.47] | 22.21 [9.36 to NA] — Insufficient number of events to calculate UL | 16.59 [4.34 to 48.20] | 18.40 [NA to NA] — Insufficient number of events to calculate LL and UL | 21.55 [10.84 to NA] — Insufficient number of events to calculate UL | 49.51 [7.72 to NA] — Insufficient number of events to calculate UL

13. Secondary Outcome: Time to Response (TTR) Assessed by Blinded Independent Central Review (BICR)
Description: Time to Response (TTR) defined as the time from randomization to the date of the first confirmed CR or PR for Cohort 3, 4 and 6, and from the first dosing date of study medication to the date of the first confirmed CR or PR for cohort 1, 2 and 5.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) to the date of attainment of complete response (CR) or partial response (PR) (up to approximately 144 months)
Population: as for outcome 12
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 3 | 2 | 2 | 11 | 8 | 10 | 7 | 8 | 4 | 16 | 16 | 15 | 3 | 5 | 10
Months | 1.41 [1.4 to 2.8] | 3.15 [2.3 to 4.0] | 1.99 [1.3 to 2.7] | 2.73 [1.3 to 6.8] | 3.63 [2.6 to 5.7] | 2.78 [1.2 to 7.0] | 1.38 [1.2 to 6.8] | 3.50 [1.9 to 5.7] | 2.81 [1.9 to 5.5] | 2.00 [1.1 to 12.8] | 2.58 [1.2 to 5.5] | 2.66 [1.2 to 8.7] | 2.66 [1.4 to 4.2] | 5.13 [1.3 to 5.7] | 4.17 [1.3 to 8.1]

14. Secondary Outcome: Time to Progression (TTP) Assessed by Blinded Independent Central Review (BICR)
Description: Time to Progression (TTP) is defined from the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) to the date of the first objectively documented disease progression. Participants who have not progressed as assessed by radiography will be censored at the last tumor assessment date prior to subsequent anti-cancer therapy. Participants who have no on-study tumor assessments were censored at the date of randomization.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) up to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (Up to approximately 144 months)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Months | 2.66 [1.38 to 4.21] | 8.21 [1.31 to NA] — Insufficient number of events to calculate UL | 2.96 [1.25 to 6.97] | 4.01 [2.76 to 4.63] | 2.79 [1.48 to 5.59] | 3.94 [2.63 to 8.05] | 2.63 [1.38 to 4.04] | 4.83 [1.94 to 5.55] | 4.63 [3.32 to 12.94] | 4.27 [2.63 to 9.69] | 1.68 [1.35 to 13.90] | 2.73 [1.45 to 5.65] | 2.79 [1.41 to 5.36] | 5.42 [2.76 to 11.47] | 11.63 [4.11 to 36.86]

15. Secondary Outcome: Time to Progression (TTP) Rate Assessed by Blinded Independent Central Review (BICR)
Description: TTP rate is defined as the percentage of participants without disease progression at select time points (milestones) during the study.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: At 6 and 12 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Percent of Participants
  6 Months | 28.6 [11.7 to 48.2] | 60.0 [25.3 to 82.7] | 27.9 [7.1 to 54.1] | 33.9 [21.4 to 46.9] | 32.8 [20.2 to 46.0] | 41.5 [26.9 to 55.5] | 26.0 [14.7 to 38.9] | 30.1 [17.3 to 44.0] | 42.5 [27.2 to 56.9] | 42.5 [28.0 to 56.3] | 43.6 [28.7 to 57.5] | 32.4 [19.3 to 46.2] | 31.6 [16.9 to 47.4] | 42.8 [25.2 to 59.3] | 50.0 [30.3 to 66.9]
  12 Months | 17.1 [4.6 to 36.5] | 24.0 [3.8 to 53.7] | 18.6 [3.0 to 44.5] | 21.4 [11.3 to 33.6] | 19.3 [9.0 to 32.4] | 30.9 [17.7 to 45.1] | 13.0 [5.3 to 24.2] | 12.2 [4.1 to 25.0] | 35.4 [20.5 to 50.6] | 33.1 [19.8 to 46.9] | 35.9 [21.9 to 50.1] | 27.6 [15.4 to 41.3] | 14.7 [4.4 to 31.0] | 32.1 [16.5 to 48.9] | 45.0 [25.5 to 62.7]

16. Secondary Outcome: Progression Free Survival (PFS) Assessed by Blinded Independent Central Review (BICR)
Description: PFS is defined as the time from randomization date or first dosing date of study medication to the date of the first objectively documented tumor progression or death due to any cause. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last tumor assessment.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm (Note: The appearance of 1or more new lesions is also considered progression).
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) up to documented disease progression or death, whichever occurs first (up to approximately 144 months)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Months | 2.69 [1.38 to 4.21] | 8.97 [1.31 to 14.06] | 2.96 [1.25 to 4.07] | 4.01 [2.76 to 4.60] | 2.76 [1.48 to 4.40] | 3.94 [2.63 to 7.23] | 2.63 [1.35 to 4.04] | 3.78 [1.84 to 5.45] | 3.91 [3.32 to 5.65] | 3.91 [2.60 to 8.31] | 1.61 [1.35 to 6.93] | 2.63 [1.31 to 4.50] | 2.30 [1.41 to 3.42] | 5.13 [2.76 to 10.91] | 4.27 [3.58 to 11.86]

17. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization date or first dosing date of study medication to the date of death (due to any cause). Participants who were alive were censored at the last known alive dates.
Time Frame: From the date of randomization (Cohort 3, 4, 6) or the date of first dose (Cohort 1, 2, 5) up to the date of death or date last known alive (up to approximately 144 months)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Months | 14.32 [5.65 to 18.14] | 36.27 [3.61 to 55.10] | 10.45 [3.68 to 20.21] | 26.68 [17.71 to 34.40] | 13.44 [8.57 to 18.89] | 17.45 [13.04 to 25.66] | 15.64 [9.69 to 20.67] | 15.24 [11.07 to 22.90] | 13.96 [8.71 to 19.25] | 22.24 [9.43 to 54.83] | 12.48 [7.62 to 16.39] | 12.75 [7.43 to 30.52] | 7.85 [4.37 to 10.51] | 20.21 [13.11 to 32.20] | 22.11 [15.15 to 36.50]

18. Secondary Outcome: Overall Survival (OS) Rate
Description: OS rate is defined as the percentage of participants who are still alive at certain time points during the study.
Time Frame: At 6, 12, 24, 48 and 60 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4 | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
Number analyzed (Participants) | 23 | 10 | 15 | 56 | 57 | 50 | 51 | 61 | 66 | 50 | 49 | 49 | 49 | 36 | 35
Percent of Participants
  6 Months | 69.6 [46.6 to 84.2] | 80.0 [40.9 to 94.6] | 53.3 [26.3 to 74.4] | 89.0 [77.0 to 94.9] | 75.4 [62.1 to 84.7] | 83.3 [69.3 to 91.3] | 84.3 [71.1 to 91.8] | 81.3 [68.8 to 89.2] | 76.7 [63.8 to 85.5] | 81.7 [67.7 to 90.0] | 75.0 [60.2 to 85.0] | 73.5 [58.7 to 83.6] | 59.2 [44.2 to 71.4] | 82.4 [64.9 to 91.7] | 82.4 [65.0 to 91.7]
  12 Months | 60.9 [38.3 to 77.4] | 80.0 [40.9 to 94.6] | 46.7 [21.2 to 68.7] | 76.0 [62.3 to 85.3] | 54.4 [40.7 to 66.2] | 67.5 [51.9 to 79.0] | 58.8 [44.1 to 70.9] | 57.1 [43.4 to 68.6] | 57.0 [43.2 to 68.6] | 60.7 [45.6 to 72.9] | 56.1 [41.0 to 68.8] | 50.8 [36.1 to 63.7] | 34.7 [21.8 to 47.9] | 70.2 [51.6 to 82.7] | 70.6 [52.3 to 83.0]
  24 Months | 26.1 [10.6 to 44.7] | 60.0 [25.3 to 82.7] | 26.7 [8.3 to 49.6] | 57.0 [42.7 to 69.0] | 26.3 [15.7 to 38.1] | 38.9 [24.5 to 53.0] | 36.6 [23.6 to 49.7] | 32.9 [21.3 to 45.0] | 30.4 [18.8 to 42.8] | 46.1 [31.7 to 59.3] | 30.2 [17.9 to 43.5] | 42.3 [28.3 to 55.7] | 10.2 [3.7 to 20.5] | 39.0 [22.6 to 55.2] | 46.1 [28.7 to 61.8]
  48 Months | 17.4 [5.4 to 35.0] | 30.0 [7.1 to 57.8] | 6.7 [0.4 to 26.0] | 20.9 [11.2 to 32.7] | 11.7 [4.9 to 21.7] | 14.6 [6.0 to 26.9] | 12.2 [5.0 to 22.9] | 15.6 [7.5 to 26.5] | 8.4 [2.7 to 18.0] | 37.0 [23.5 to 50.6] | 21.6 [11.2 to 34.2] | 25.4 [14.2 to 38.2] | 00 [00 to 00] | 19.0 [7.5 to 34.4] | 30.7 [16.1 to 46.6]
  60 Months | 8.7 [1.5 to 24.2] | 15.0 [1.0 to 45.7] | 6.7 [0.4 to 26.0] | 15.2 [7.1 to 26.1] | 9.7 [3.7 to 19.3] | 14.6 [6.0 to 26.9] | 12.2 [5.0 to 22.9] | 8.9 [3.0 to 18.8] | 5.6 [1.2 to 15.1] | 29.6 [17.1 to 43.2] | 19.2 [9.4 to 31.6] | 21.2 [11.0 to 33.6] | 00 [00 to 00] | 15.2 [5.1 to 30.2] | 24.6 [11.6 to 40.0]

19. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Cmax is the maximum observed serum concentration.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: All treated participants in Cohort 1 with baseline and at least 1 post-baseline assessment; uninfected HCC, HCV-infected, and HBV-infected participants reported together as pre-specified.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 23 | 10 | 15
ug/mL
  Cycle 1 Day 1 | 60.06 (335.87) | 19.81 (109.88) | 9.82 (244.81)
  Cycle 3 Day 1: number analyzed (Participants) | 8 | 6 | 3
  Cycle 3 Day 1 | 100.74 (339.27) | 23.09 (130.66) | 15.54 (379.81)

20. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Tmax is the time taken to reach the maximum observed serum concentration (Cmax).
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Median (Full Range); unit: Hour
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 23 | 10 | 15
Hour
  Cycle 1 Day 1 | 3.00 [1.0 to 25.2] | 2.98 [0.9 to 25.2] | 3.00 [0.9 to 23.9]
  Cycle 3 Day 1: number analyzed (Participants) | 8 | 6 | 3
  Cycle 3 Day 1 | 12.75 [0.9 to 24.3] | 12.28 [1.0 to 24.5] | 24.13 [0.8 to 25.7]

21. Secondary Outcome: Area Under the Serum Concentration Time Curve in the Dosing Interval [AUC(TAU)]
Description: AUC (TAU) is the area measured under the concentration-time curve taken over the dosing interval.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug.h/mL
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 21 | 9 | 15
ug.h/mL
  Cycle 1 Day 1 | 9114.43 (366.71) | 2825.09 (159.47) | 1313.76 (287.76)
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 5 | 3
  Cycle 3 Day 1 | 15229.27 (383.94) | 3358.78 (79.68) | 3731.16 (505.00)

22. Secondary Outcome: Serum Concentration Achieved at the End of Dosing Interval (Trough Concentration) (Ctrough)
Description: Ctrough is the lowest observed serum concentration.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 21 | 9 | 15
ug/mL
  Cycle 1 Day 1 | 16.52 (383.95) | 4.40 (194.65) | 2.26 (412.75)
  Cycle 3 Day 1: number analyzed (Participants) | 6 | 5 | 3
  Cycle 3 Day 1 | 32.48 (430.86) | 6.76 (97.21) | 8.51 (473.58)

23. Secondary Outcome: Serum Concentration Achieved at the End of the Infusion (Ceoinf)
Description: Serum Concentration Achieved at the End of the Infusion (Ceoinf) refers to the amount of drug present in the blood (serum) immediately after the completion of an infusion. It represents the concentration measured at the exact time the infusion ends, before any significant elimination or distribution occurs.
Time Frame: At Cycle 1 Day 1 and Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 23 | 10 | 14
ug/mL
  Cycle 1 Day 1 | 49.88 (315.39) | 17.07 (123.95) | 6.99 (254.53)
  Cycle 3 Day 1: number analyzed (Participants) | 8 | 5 | 5
  Cycle 3 Day 1 | 84.36 (371.92) | 25.53 (147.16) | 11.80 (353.06)

24. Secondary Outcome: Ratio of an Exposure Measure at Steady State to That After the First Dose (Exposure Measure Includes Cmax) (AI_Cmax)
Description: AI_Cmax is ratio of an exposure measure at steady state to that after the first dose (exposure measure includes Cmax)
Time Frame: At Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 8 | 6 | 3
Ratio | 2.26 (69.85) | 1.53 (23.34) | 1.45 (23.94)

25. Secondary Outcome: Accumulation Index Ratio of AUC at Steady State to That After the First Dose (AI_AUC)
Description: AI_AUC is accumulation index ratio of AUC at steady state to that after the first dose
Time Frame: At Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 6 | 5 | 3
Ratio | 2.60 (24.54) | 2.23 (9.80) | 2.28 (8.90)

26. Secondary Outcome: Effective T-Half (T-HALF)
Description: Effective half-life is defined as the time it takes for the amount of a drug in the body to decrease by half.
Time Frame: At Cycle 3 Day 1 (Each Cycle = 2 Weeks)
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Cohort 1 Uninfected HCC | Cohort 1 HCV Infected | Cohort 1 HBV Infected
Number analyzed (Participants) | 6 | 5 | 3
Hour | 468.07 (27.65) | 382.36 (15.52) | 406.60 (15.65)

27. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: Baseline ADA Positive: Participant with baseline ADA-positive sample ADA Positive: Participant with at least one ADA-positive sample relative to baseline Persistent Positive (PP): ADA-positive sample at 2 or more consecutive timepoints Not PP-Last Sample Positive: Not persistent but with ADA-positive sample at the last sampling timepoint Other Positive: Not persistent but some ADA-positive samples with the last sample being negative ADA Negative: Participant with no ADA-positive sample after initiation of treatment
Time Frame: as for outcome 1
Population: All treated participants in Cohort 1 and 2 with baseline and at least 1 post-baseline assessment. Pre-specified to be reported for Cohort 1 and 2 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2 Uninfected Sorafenib Naive/Intolerant: Treatment 1 | Cohort 2 Uninfected Sorafenib Progressors: Treatment 2 | Cohort 2 HCV Infected: Treatment 3 | Cohort 2 HBV Infected: Treatment 4
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 12 | 3 | 4 | 3 | 5 | 3 | 3 | 4 | 53 | 54 | 44 | 50
Participants
  Baseline ADA Positive | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 3 | 5 | 1
  ADA Positive | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 18 | 19 | 16 | 7
  ADA Positive [Persistent Positive (PP)] | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 3 | 0
  ADA Positive [Not PP-Last Sample Positive] | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 3 | 9 | 1
  ADA Positive [Other Positive] | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 12 | 15 | 4 | 6
  Neutralizing Positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  ADA Negative | 1 | 1 | 1 | 3 | 11 | 1 | 3 | 3 | 4 | 2 | 2 | 3 | 35 | 35 | 28 | 43

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from the date of their randomization (Cohorts 3, 4, and 6) or first dose (Cohorts 1, 2, and 5) until study completion (assessed up to approximately 144 months). SAEs and Other AEs were assessed from first dose of study medication through 100 days following last dose of study treatment (Assessed for approximately 04 months up to a max of approximately 106 months).
Description: The number at Risk for All-Cause Mortality represents all randomized participants (Cohorts 3, 4, and 6) or all participants that received at lease 1 dose of study medication (Cohorts 1, 2, and 5).
  Serious Adverse Events and Other (Not Including Serious) Adverse Events represent all participants that received at least 1 dose of study medication.
  Additionally, Cohort 2 participants were pre-specified to be reported together.
Groups:
- Cohort 2: Nivolumab 3 mg/kg: Participants received nivolumab 3 mg/kg every 2 weeks
Arm/Group | Cohort 1 Uninfected HCC: Treatment 1 | Cohort 1 Uninfected HCC: Treatment 2 | Cohort 1 Uninfected HCC: Treatment 3 | Cohort 1 Uninfected HCC: Treatment 4 | Cohort 1 Uninfected HCC: Treatment 5 | Cohort 1 HCV Infected: Treatment 6 | Cohort 1 HCV Infected: Treatment 7 | Cohort 1 HCV Infected: Treatment 8 | Cohort 1 HBV Infected: Treatment 9 | Cohort 1 HBV Infected: Treatment 10 | Cohort 1 HBV Infected: Treatment 11 | Cohort 1 HBV Infected: Treatment 12 | Cohort 2: Nivolumab 3 mg/kg | Cohort 3: Treatment 1 | Cohort 3: Treatment 2 | Cohort 4: Treatment 1 | Cohort 4: Treatment 2 | Cohort 4: Treatment 3 | Cohort 5: Treatment 1 | Cohort 6: Treatment 1 | Cohort 6: Treatment 2
All-Cause Mortality (participants affected / at risk) | 1/1 | 3/3 | 2/3 | 2/3 | 13/13 | 1/3 | 4/4 | 3/3 | 5/5 | 3/3 | 3/3 | 4/4 | 186/214 | 52/61 | 53/66 | 36/50 | 41/49 | 41/49 | 48/49 | 29/36 | 26/35
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 2/3 | 0/3 | 8/13 | 0/3 | 3/4 | 1/3 | 5/5 | 3/3 | 1/3 | 3/4 | 137/214 | 35/60 | 33/62 | 35/49 | 36/49 | 36/48 | 37/49 | 22/36 | 25/35
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 3/3 | 3/3 | 13/13 | 3/3 | 4/4 | 3/3 | 5/5 | 3/3 | 3/3 | 4/4 | 210/214 | 55/60 | 57/62 | 47/49 | 47/49 | 45/48 | 42/49 | 36/36 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Uninfected HCC: Treatment 1 (N=1) | Cohort 1 Uninfected HCC: Treatment 2 (N=3) | Cohort 1 Uninfected HCC: Treatment 3 (N=3) | Cohort 1 Uninfected HCC: Treatment 4 (N=3) | Cohort 1 Uninfected HCC: Treatment 5 (N=13) | Cohort 1 HCV Infected: Treatment 6 (N=3) | Cohort 1 HCV Infected: Treatment 7 (N=4) | Cohort 1 HCV Infected: Treatment 8 (N=3) | Cohort 1 HBV Infected: Treatment 9 (N=5) | Cohort 1 HBV Infected: Treatment 10 (N=3) | Cohort 1 HBV Infected: Treatment 11 (N=3) | Cohort 1 HBV Infected: Treatment 12 (N=4) | Cohort 2: Nivolumab 3 mg/kg (N=214) | Cohort 3: Treatment 1 (N=60) | Cohort 3: Treatment 2 (N=62) | Cohort 4: Treatment 1 (N=49) | Cohort 4: Treatment 2 (N=49) | Cohort 4: Treatment 3 (N=48) | Cohort 5: Treatment 1 (N=49) | Cohort 6: Treatment 1 (N=36) | Cohort 6: Treatment 2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 3 | 3 | 2 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3 | 3 | 1 | 2 | 2 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 1 | 6 | 2 | 1 | 3 | 3 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune enteropathy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0 | 1 | 0 | 2 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 0 | 3 | 1 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 2 | 2 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hernia pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7 | 2 | 0 | 4 | 3 | 4 | 0 | 3 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Type IV hypersensitivity reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleurisy bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1 | 0 | 2 | 3 | 0 | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spontaneous bacterial peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 1 | 3 | 3 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 6 | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inflammatory marker increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 2
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 0 | 1 | 2 | 0 | 3 | 52 | 10 | 10 | 12 | 15 | 18 | 18 | 6 | 5
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bell's palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial tumour haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Quadriplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Loss of personal independence in daily activities (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Uninfected HCC: Treatment 1 (N=1) | Cohort 1 Uninfected HCC: Treatment 2 (N=3) | Cohort 1 Uninfected HCC: Treatment 3 (N=3) | Cohort 1 Uninfected HCC: Treatment 4 (N=3) | Cohort 1 Uninfected HCC: Treatment 5 (N=13) | Cohort 1 HCV Infected: Treatment 6 (N=3) | Cohort 1 HCV Infected: Treatment 7 (N=4) | Cohort 1 HCV Infected: Treatment 8 (N=3) | Cohort 1 HBV Infected: Treatment 9 (N=5) | Cohort 1 HBV Infected: Treatment 10 (N=3) | Cohort 1 HBV Infected: Treatment 11 (N=3) | Cohort 1 HBV Infected: Treatment 12 (N=4) | Cohort 2: Nivolumab 3 mg/kg (N=214) | Cohort 3: Treatment 1 (N=60) | Cohort 3: Treatment 2 (N=62) | Cohort 4: Treatment 1 (N=49) | Cohort 4: Treatment 2 (N=49) | Cohort 4: Treatment 3 (N=48) | Cohort 5: Treatment 1 (N=49) | Cohort 6: Treatment 1 (N=36) | Cohort 6: Treatment 2 (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 42 | 5 | 8 | 6 | 11 | 11 | 8 | 6 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 1 | 3 | 1 | 2 | 2 | 3 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 3
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 4 | 0 | 1 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 3 | 3 | 1 | 2 | 4
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 10 | 3 | 0 | 11 | 5 | 6 | 1 | 7 | 5
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 0
Pterygium (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 1 | 3 | 2 | 2 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 30 | 7 | 1 | 4 | 3 | 6 | 4 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 51 | 14 | 14 | 7 | 15 | 7 | 7 | 4 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 24 | 7 | 4 | 8 | 5 | 4 | 2 | 2 | 3
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 22 | 6 | 10 | 8 | 6 | 8 | 18 | 6 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 40 | 11 | 10 | 9 | 11 | 12 | 2 | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 4 | 3 | 1 | 0 | 1 | 1 | 2 | 2 | 61 | 11 | 32 | 19 | 11 | 19 | 9 | 21 | 15
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 23 | 2 | 4 | 6 | 4 | 3 | 0 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 13 | 2 | 1 | 6 | 4 | 3 | 1 | 2 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 3 | 2 | 0 | 4 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 43 | 10 | 13 | 10 | 13 | 11 | 2 | 5 | 5
Neurogenic bowel (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 11 | 3 | 5 | 6 | 3 | 3 | 2 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 37 | 8 | 6 | 6 | 10 | 7 | 0 | 5 | 7
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 5 | 6 | 5 | 6 | 5 | 7 | 6 | 7
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 2 | 5 | 0 | 2 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 5 | 1 | 3 | 0 | 2 | 1 | 0 | 1 | 86 | 23 | 21 | 11 | 11 | 13 | 5 | 10 | 11
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 19 | 1 | 1 | 7 | 6 | 5 | 0 | 1 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 13 | 0 | 1 | 7 | 5 | 6 | 2 | 1 | 3
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 4 | 1 | 1 | 0 | 0 | 3 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 35 | 8 | 7 | 10 | 11 | 14 | 13 | 4 | 7
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 3 | 1 | 1 | 1 | 3 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 40 | 15 | 11 | 14 | 15 | 19 | 8 | 10 | 9
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 2 | 3 | 3 | 5
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 1 | 5 | 2 | 2 | 1 | 2 | 4
Nasal herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 2 | 3 | 2 | 2 | 1 | 5 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 4 | 0 | 2 | 1 | 1 | 1
Pustule (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 3 | 1 | 0 | 0 | 13 | 2 | 1 | 1 | 6 | 2 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 10 | 2 | 1 | 1 | 1 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 0 | 4 | 0 | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 36 | 9 | 7 | 15 | 11 | 9 | 2 | 6 | 15
Amylase increased (Investigations) | 0 | 0 | 2 | 2 | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 0 | 20 | 2 | 3 | 5 | 5 | 4 | 4 | 1 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 4 | 2 | 2 | 0 | 2 | 0 | 1 | 1 | 38 | 10 | 10 | 17 | 16 | 11 | 6 | 10 | 15
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 12 | 3 | 5 | 6 | 3 | 5 | 0 | 3 | 6
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 19 | 7 | 7 | 10 | 7 | 2 | 6 | 5 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 6 | 3 | 0 | 4 | 1 | 0 | 2 | 3 | 1
Cortisol decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 5 | 2 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 2 | 0 | 0 | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 18 | 3 | 4 | 9 | 7 | 9 | 5 | 4 | 9
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 1 | 3 | 4 | 3 | 1 | 2 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 13 | 3 | 4 | 10 | 3 | 0 | 1 | 4 | 7
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 5 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 17 | 2 | 11 | 11 | 6 | 5 | 0 | 5 | 6
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 3 | 2 | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 3 | 0 | 2 | 2 | 2 | 3 | 57 | 12 | 22 | 20 | 13 | 15 | 2 | 8 | 8
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 1 | 1 | 1 | 3 | 4 | 2 | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 15 | 6 | 4 | 3 | 3 | 6 | 1 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 3 | 1 | 4 | 2 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 15 | 5 | 5 | 5 | 2 | 5 | 1 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6 | 2 | 3 | 4 | 5 | 6 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9 | 2 | 3 | 1 | 1 | 3 | 1 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 2 | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 7 | 8 | 3 | 9 | 4 | 6 | 2 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 13 | 1 | 8 | 3 | 0 | 2 | 0 | 3 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 38 | 5 | 5 | 9 | 10 | 7 | 4 | 6 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 2 | 1 | 1 | 0 | 0 | 2 | 37 | 9 | 10 | 8 | 3 | 10 | 2 | 4 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 3
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 2 | 1 | 1 | 1 | 3 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 3 | 2 | 4 | 4 | 0 | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 2 | 6 | 9 | 3 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 14 | 2 | 7 | 9 | 3 | 4 | 1 | 1 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 25 | 3 | 3 | 9 | 5 | 7 | 1 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4 | 4 | 2 | 1 | 2 | 1 | 5 | 3 | 6
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 23 | 5 | 6 | 11 | 2 | 5 | 2 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 2 | 1 | 3 | 2 | 2 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 12 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 4 | 3 | 0 | 2 | 2 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 27 | 5 | 5 | 11 | 5 | 9 | 2 | 2 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 3 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 3 | 1 | 0 | 0 | 54 | 7 | 6 | 20 | 12 | 9 | 5 | 4 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 9 | 0 | 0 | 0 | 1 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 19 | 7 | 5 | 7 | 8 | 9 | 1 | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 4 | 2 | 2 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 2 | 3 | 1 | 2 | 0 | 3 | 2
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 6 | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 1 | 4 | 4 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 1 | 14 | 0 | 0 | 5 | 1 | 1 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 14 | 3 | 8 | 4 | 3 | 2 | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 0 | 1 | 1 | 1 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 8 | 29 | 2 | 1 | 0 | 0 | 13 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 6 | 2 | 1 | 0 | 2 | 1 | 0 | 1 | 71 | 13 | 7 | 27 | 24 | 18 | 13 | 11 | 10
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 7 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 43 | 10 | 11 | 16 | 15 | 12 | 3 | 6 | 9
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 2 | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 7 | 1 | 5 | 8 | 5 | 3 | 2 | 2 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 2 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 24 | 8 | 15 | 4 | 4 | 4 | 2 | 12 | 17
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 7 | 4 | 4 | 5 | 4 | 3 | 1 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT01658878/Prot_SAP_000.pdf